CLINICAL TRIAL: NCT02951234
Title: Kawasaki Disease Center, Kaohsiung Chang Gung Memorial Hospital, Taiwan
Brief Title: A Multi-center, Randomized to Compare the Efficacy of IVIG Alone and IVIG Plus High-dose Aspirin in Kawasaki Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVIG And Aspirin in KD
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Kawasaki Disease
Keywords: coronary artery lesions; intravenous immunoglobulin; Kawasaki disease; randomized clinical trial; aspirin
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulins, Intravenous; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG only (Experimental): All patients will receive IVIG (2g/kg) in 10-12 hours alone, without high-dose aspirin. After fever subsides, low-dose aspirin (3-5mg/kg/day) will be prescribed until 6-8 weeks.
  Interventions: Other: IVIG only
- IVIG and Aspirin (Active Comparator): All patients will receive IVIG (2g/kg) in 10-12 hours plus high-dose aspirin (80-100mg/kg/day, divided into four doses) till fever subside. After fever subsides, low-dose aspirin (3-5mg/kg/day) will be prescribed until 6-8 weeks.
  Interventions: Other: IVIG and Aspirin

INTERVENTIONS:
Other: IVIG only — All patients will receive IVIG (2g/kg) in 10-12 hours alone, without high-dose aspirin.
  Arms: IVIG only
Other: IVIG and Aspirin — All patients will receive IVIG (2g/kg) in 10-12 hours plus high-dose aspirin (80-100mg/kg/day, divided into four doses) till fever subside.
  Arms: IVIG and Aspirin

SUMMARY:
Kawasaki disease (KD) is an acute febrile systemic vasculitis most commonly seen in children under the age of 5 years old. This trial has been designed as a multi-center, prospective, randomized controlled, evaluator-blinded trial with two parallel groups to determine whether IVIG alone as the primary therapy in acute-stage KD is as effective as IVIG combined with high-dose aspirin therapy. The primary endpoint is defined as CAL formation at 6-8 weeks.

DETAILED DESCRIPTION:
Background: Kawasaki disease (KD) is an acute febrile systemic vasculitis most commonly seen in children under the age of 5 years old. High-dose aspirin is often administered, but the duration of such treatment varies. Many centers reduce the aspirin dose once the patient is afebrile, even before treating said patient with IVIG. However, a randomized controlled trial regarding high-dose aspirin in the acute stage of KD has not previously been carried out.

Methods/design: This trial has been designed as a multi-center, prospective, randomized controlled, evaluator-blinded trial with two parallel groups to determine whether IVIG alone as the primary therapy in acute-stage KD is as effective as IVIG combined with high-dose aspirin therapy. The primary endpoint is defined as CAL formation at 6-8 weeks. Patients meeting the eligibility criteria are randomly assigned (1:1) to a test group (that receives only IVIG) or a standard group (that receives IVIG plus high-dose aspirin). This clinical trial is conducted at seven medical centers in Taiwan.

Discussion: Since high-dose aspirin has significant anti-inflammatory and anti-platelet functions, it does not appear to lower the frequency of disease outcomes. Furthermore, it can decrease hemoglobin levels. Therefore, the investigators have initiated this randomized controlled trial to determine whether high-dose aspirin is necessary in the acute stage of KD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, under the age of 7 years old.

2. Fulfilled the AHA criteria for KD as explained below:

1. Fever (more than 38.0℃ ear temperature) > or = 5 days, as well as 4 of the 5 following symptoms
2. Diffuse mucosal inflammation (strawberry tongue, dry and cracked lips)
3. Bilateral non-purulent conjunctivitis
4. Dysmorphous skin rashes
5. Indurative edematous change over the hands and feet, or desquamation over the fingertips or toes
6. Cervical lymphadenopathy (one or more nodule at least 1.5 cm in diameter)

3. An informed consent form (ICF, appendix B) signed by the patient or a legal guardian.

-

Exclusion Criteria:

1. Had symptoms that did not completely match the KD criteria.
2. Had an acute fever for < 5 days and >10 days
3. IVIG treatment at another hospital before being referred to the study center.
4. Treatment with corticosteroids, other than the inhaled form, in the two weeks prior to joining the study;
5. The presence of a disease known to mimic Kawasaki disease (such as adenovirus infection, toxic shock syndrome etc.).
6. Previous KD diagnosis.
7. Inability to take aspirin (such as history of hypersensitivity to aspirin, G6PD deficiency, recent herpes zoster infection or vaccination, etc.)
8. Afebrile prior to enrollment
9. CAL prior to enrollment
10. Severe concomitant medical disorders (e.g., immunodeficiency, chromosomal anomalies, congenital heart diseases, metabolic diseases, nephritis, collagen diseases, etc.)
11. Suspected to have an infectious disease, including sepsis, septic meningitis, peritonitis, bacterial pneumonia, varicella, and influenza
12. Judged by the researcher to be unsuitable for this trial.

    -

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
coronary artery lesions | 8 weeks

SECONDARY OUTCOMES:
IVIG resistance | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Chang Kuo, MD, PhD, Principal Investigator — Kawasaki Disease Center, Kaohsiung Chang Gung Memorial Hospital
Locations (5):
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung Metroharbor Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuo HC, Lin MC, Kao CC, Weng KP, Ding Y, Han Z, Chen CJ, Jan SL, Chien KJ, Ko CH, Lin CY, Lei WT, Guo MM, Yang KD, Sylvester KG, Whitin JC, Tian L, Chubb H, Ceresnak SR, McElhinney D, Cohen HJ, Ling XB. Intravenous Immunoglobulin Alone for Coronary Artery Lesion Treatment of Kawasaki Disease: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e253063. doi: 10.1001/jamanetworkopen.2025.3063. PMID 40178858
- [Derived] Kuo HC, Lin MC, Kao CC, Weng KP, Ding Y, Chen CJ, Jan SL, Chien KJ, Ko CH, Lin CY, Lei WT, Chang LS, Guo MM, Yang KD, Sylvester KG, Han Z, Whitin JC, Tian L, Chubb H, Ceresnak SR, McElhinney D, Cohen HJ, Ling XB. EFFICACY OF INTRAVENOUS IMMUNOGLOBULIN ALONE ON CORONARY ARTERY LESION REDUCTION IN KAWASAKI DISEASE. medRxiv [Preprint]. 2024 Jul 12:2024.07.11.24310310. doi: 10.1101/2024.07.11.24310310. PMID 39040184
- [Derived] Kuo HC, Guo MM, Lo MH, Hsieh KS, Huang YH. Effectiveness of intravenous immunoglobulin alone and intravenous immunoglobulin combined with high-dose aspirin in the acute stage of Kawasaki disease: study protocol for a randomized controlled trial. BMC Pediatr. 2018 Jun 22;18(1):200. doi: 10.1186/s12887-018-1180-1. PMID 29933749